CLINICAL TRIAL: NCT01974895
Title: Immunogenicity and Safety Study of GSK Biologicals' Quadrivalent Influenza Vaccine (GSK2282512A) in Children 6 to 35 Months of Age
Brief Title: Study to Evaluate Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Quadrivalent Influenza Vaccine GSK2282512A When Administered to Children From 6 to 35 Months of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 200806
Record Dates: First submitted 2013-10-23; First posted 2013-11-04 (Estimated); Results first posted 2015-04-13 (Estimated); Last update posted 2018-09-07 (Actual); Status verified 2016-08

CONDITIONS: Influenza
Keywords: Children; Immunogenicity; Fluzone®; 6 to 35 months of age; Seasonal influenza; Safety
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor

ARMS (2):
- FluLaval Quadrivalent Group (Experimental): Subjects received 1 or 2 doses of FluLaval® Quadrivalent vaccine at Day 0 or Days 0 and 28, depending on age and vaccine priming status.
  Interventions: Biological: FluLaval® Quadrivalent
- Fluzone Group (Active Comparator): Subjects received 1 or 2 doses of Fluzone® vaccine at Day 0 or Days 0 and 28, depending on age and priming status.
  Interventions: Biological: Fluzone®

INTERVENTIONS:
Biological: FluLaval® Quadrivalent — 1 or 2 doses administered intramuscularly (IM) in deltoid region of non-dominant arm (for subjects ≥12 months of age) or anterolateral region of left thigh (for subjects <12 months of age) on Day 0 (primed subjects) and on Day 0 and Day 28 (unprimed subjects), respectively.
  Other Names: GSK2282512A
  Arms: FluLaval Quadrivalent Group
Biological: Fluzone® — 1 or 2 doses administered IM in deltoid region of non-dominant arm (for subjects ≥12 months of age) or anterolateral region of left thigh (for subjects <12 months of age) on Day 0 (primed subjects) and on Day 0 and Day 28 (unprimed subjects), respectively.
  Arms: Fluzone Group

SUMMARY:
The purpose of this study is to evaluate the immunogenicity and safety of the new influenza vaccine GSK2282512A (FLU Q-QIV) and compare its activity to Sanofi Pasteur's Fluzone® (TIV) in children 6 to 35 months of age.

DETAILED DESCRIPTION:
The subjects will be randomised (1:1) in the two treatment groups (Q-QIV and TIV-YB) to explore response to vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Subjects' parent(s)/Legally Acceptable Representative(s) [LAR(s)] who, in the opinion of the investigator, can and will comply, with the requirements of the protocol.
* A male or female between, and including, 6 and 35 months of age at the time of the first vaccination.
* Written informed consent obtained from the parent(s)/LAR(s) of the subject.
* Subjects in stable health as determined by investigator's clinical examination and assessment of subject's medical history.
* Subjects are eligible regardless of history of administration of influenza vaccine in a previous season.

Exclusion Criteria:

* Use of any investigational or non-registered product other than the study vaccine within 30 days preceding the first dose of study vaccine, or planned use during the study period. Routine registered childhood vaccinations are permitted.
* Child in care.
* Chronic administration of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose. For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, or equivalent. Inhaled and topical steroids are allowed.
* Prior receipt of any seasonal or pandemic influenza vaccine within six months preceding the first dose of study vaccine, or planned use during the study period.
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.
* History of Guillain-Barré syndrome within six weeks of receipt of prior influenza vaccine.
* Any known or suspected allergy to any constituent of influenza vaccines; a history of anaphylactic-type reaction to consumption of eggs; or a history of severe adverse reaction to a previous influenza vaccine.
* Acute disease and/or fever at the time of enrollment.

  * Fever is defined as temperature ≥ 38.0°C/100.4°F by any method.
  * Subjects with a minor illness without fever may be enrolled at the discretion of the investigator.
* Any significant disorder of coagulation or treatment with warfarin derivatives or heparin.
* Any confirmed or suspected immunosuppressive or immunodeficient condition, based on medical history and physical examination.
* Any other condition which, in the opinion of the investigator, prevents the subject from participating in the study.

Ages: 6 Months to 35 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 316 (Actual)
Dates: Start 2013-10-23; Primary Completion 2014-02-27 (Actual); Study Completion 2014-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (12):
  - GSK Investigational Site, Sacramento, California
  - GSK Investigational Site, West Covina, California
  - GSK Investigational Site, Altamonte Springs, Florida
  - GSK Investigational Site, Fall River, Massachusetts
  - GSK Investigational Site, Woburn, Massachusetts
  - GSK Investigational Site, Stevensville, Michigan
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Hermitage, Pennsylvania
  - GSK Investigational Site, Barnwell, South Carolina
  - GSK Investigational Site, Cheraw, South Carolina
  - GSK Investigational Site, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 200806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 200806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 200806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 200806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 200806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 200806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 200806 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Not all subjects who withdrew from the study were willing to provide a reason for withdrawal. Thus, the reasons for withdrawal for these subjects are unknown.
Pre-assignment Details: 2 subjects were allocated subject numbers but study vaccine was not administered, thus were excluded from the study prior to group assignment.
Period: Overall Study
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Started | 158 | 156
Completed | 143 | 141
Not Completed | 15 | 15
Not completed — Protocol Violation | 1 | 0
Not completed — Lost to Follow-up | 4 | 6
Not completed — Withdrawal by Subject | 0 | 1
Not completed — Other (Missed Visit) | 1 | 0
Not completed — Other (Reason unknown) | 9 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group | Total
Number analyzed (Participants) | 158 | 156 | 314
Age, Continuous [Mean (Standard Deviation); unit: Months] | 19.6 (8.8) | 19.8 (8.9) | 19.7 (8.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 82 | 156
  Male | 84 | 74 | 158

OUTCOME MEASURES:

1. Primary Outcome: Number of Seroconverted Subjects for Haemagglutination Inhibition (HI) Antibodies Against Each of the Four Vaccine Influenza Strains of FluLaval® Quadrivalent Vaccine.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
  The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/2/2012 (Yamagata), Flu B/Brisbane/60/2008 (Victoria). This outcome concerns solely subjects in the FluLaval Quadrivalent Group.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: 28 days after the last vaccine dose (at Day 28 for primed subjects and at Day 56 for unprimed subjects)
Population: Analysis was performed on the According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 143 | 137
Subjects
  H1N1 [Day 28 = primed and Day 56 = unprimed] | 115 | NA — This primary outcome concerns solely subjects in the FluLaval Quadrivalent Group.
  H3N2 [Day 28 = primed and Day 56 = unprimed] | 103 | NA — This primary outcome concerns solely subjects in the FluLaval Quadrivalent Group.
  Yamagata [Day 28 = primed and Day 56 = unprimed] | 123 | NA — This primary outcome concerns solely subjects in the FluLaval Quadrivalent Group.
  Victoria [Day 28 = primed and Day 56 = unprimed] | 95 | NA — This primary outcome concerns solely subjects in the FluLaval Quadrivalent Group.

2. Secondary Outcome: Number of Seroconverted Subjects for HI Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: A seroconverted subject was defined as a vaccinated subject with either a pre-vaccination titer less than (<) 1:10 and a post-vaccination titer greater than or equal to (≥) 1:40, or a pre-vaccination titer ≥ 1:10 and at least a 4-fold increase in post-vaccination titer.
  The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/2/2012 (Yamagata), Flu B/Brisbane/60/2008 (Victoria). This outcome concerns solely subjects in the Fluzone Group.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: 28 days after the last vaccine dose (at Day 28 for primed subjects and at Day 56 for unprimed subjects)
Population: Analysis was performed on the ATP cohort for immunogenicity which included all evaluable subjects for whom data concerning immunogenicity outcome measures were available and subjects for whom assay results were available for antibodies against at least one study vaccine antigen component after vaccination.
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 143 | 137
Subjects
  H1N1, [Day 28 = primed and Day 56 = unprimed] | NA — This outcome concerns solely subjects in the Fluzone Group. | 98
  H3N2, [Day 28 = primed and Day 56 = unprimed] | NA — This outcome concerns solely subjects in the Fluzone Group. | 94
  Yamagata, [Day 28 = primed and Day 56 = unprimed] | NA — This outcome concerns solely subjects in the Fluzone Group. | 115
  Victoria, [Day 28 = primed and Day 56 = unprimed] | NA — This outcome concerns solely subjects in the Fluzone Group. | 17

3. Secondary Outcome: Haemagglutination Inhibition (HI) Antibody Titers Against Each of the Four Vaccine Influenza Strains
Description: HI antibody titres were expressed as Geometric mean titers (GMTs). The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/2/2012 (Yamagata), Flu B/Brisbane/60/2008 (Victoria).
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: On Day 0 and 28 days after the last vaccine (Day 28 and Day 56 for primed and unprimed subjects respectively)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 143 | 137
Titers
  H1N1, [Day 0] | 10.3 [8.6 to 12.3] | 10.0 [8.3 to 11.9]
  H1N1, [Day 28 = primed and Day 56 = unprimed] | 141.3 [115.1 to 173.5] | 90.8 [73.2 to 112.6]
  H3N2, [Day 0] | 11.1 [9.1 to 13.5] | 11.5 [9.3 to 14.2]
  H3N2, [Day 28 = primed and Day 56 = unprimed] | 100.6 [82.6 to 122.6] | 86.2 [70.6 to 105.4]
  Yamagata, [Day 0] | 14.5 [12.1 to 17.5] | 12.3 [10.3 to 14.7]
  Yamagata, [Day 28 = primed and Day 56 = unprimed] | 212.0 [174.6 to 257.3] | 140.0 [113.9 to 172.0]
  Victoria, [Day 0] | 7.7 [6.6 to 9.1] | 6.6 [5.9 to 7.5]
  Victoria, [Day 28 = primed and Day 56 = unprimed] | 69.0 [54.9 to 86.6] | 12.8 [10.6 to 15.4]

4. Secondary Outcome: Number of Subjects Who Were Seroprotected for HI Antibodies Against Each of the Four Vaccine Influenza Strains.
Description: A seroprotected subject was defined as a vaccinated subject with a serum HI titer greater than or equal to (≥) 1:40 that usually is accepted as indicating protection in adults. The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/2/2012 (Yamagata), Flu B/Brisbane/60/2008 (Victoria).
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: At Day 0 (for all subjects) and Day 28 after last vaccine dose (Day 28 for primed subjects and Day 56 for unprimed subjects)
Population: as for outcome 2
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 143 | 137
Subjects
  H1N1, [Day 0] | 25 | 22
  H1N1, [Day 28 = primed and Day 56 = unprimed] | 125 | 111
  H3N2, [Day 0] | 29 | 25
  H3N2, [Day 28 = primed and Day 56 = unprimed] | 118 | 110
  Yamagata, [Day 0] | 31 | 22
  Yamagata, [Day 28 = primed and Day 56 = unprimed] | 135 | 124
  Victoria, [Day 0] | 13 | 9
  Victoria, [Day 28 = primed and Day 56 = unprimed] | 101 | 27

5. Secondary Outcome: Mean Geometric Increase (MGI) for HI Antibody Titer Against Each of the Four Vaccine Influenza Strains.
Description: MGI was defined as the fold increase in serum haemagglutination inhibition (HI) GMTs post-vaccination compared to pre-vaccination (Day 0). The vaccine strains assessed were Flu A/California/7/2009 (H1N1), Flu A/Texas/50/2012 (H3N2), Flu B/Massachusetts/2/2012 (Yamagata), Flu B/Brisbane/60/2008 (Victoria).
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: 28 days after the last vaccine dose (at Day 28 for primed subjects and at Day 56 for unprimed subjects)
Population: as for outcome 2
Measure: Geometric Mean (95% Confidence Interval); unit: Fold increase
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 143 | 137
Fold increase
  H1N1, [Day 28 = primed and Day 56 = unprimed] | 13.73 [11.10 to 16.99] | 9.11 [7.32 to 11.33]
  H3N2, [Day 28 = primed and Day 56 = unprimed] | 9.09 [7.69 to 10.76] | 7.53 [6.36 to 8.90]
  Yamagata, [Day 28 = primed and Day 56 = unprimed] | 14.59 [11.72 to 18.16] | 11.36 [9.09 to 14.19]
  Victoria, [Day 28 = primed and Day 56 = unprimed] | 8.94 [7.34 to 10.89] | 1.93 [1.69 to 2.19]

6. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Symptoms.
Description: Solicited local symptoms assessed were pain, redness and swelling. Any was defined as occurrence of the specified solicited local symptom regardless of its intensity. Grade 3 pain was defined as pain that made the subject cry when limb was moved/spontaneously painful. Grade 3 swelling was greater than 100 millimeters (mm) i.e. >100mm.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: During a 7-day follow-up period (i.e. day of vaccination and six subsequent days) after each vaccination
Population: Analysis was performed on the Total Vaccinated cohort, which included all subjects with vaccine administration documented and for whom safety data were available.
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 151 | 148
Subjects
  Any Pain | 48 | 48
  Grade 3 Pain | 4 | 1
  Any Redness | 2 | 0
  Grade 3 Redness | 0 | 0
  Any Swelling | 0 | 1
  Grade 3 Swelling | 0 | 0

7. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General Symptoms.
Description: Solicited general symptoms assessed were drowsiness, irritability/fussiness and loss of appetite. Any was defined as any solicited general symptom reported irrespective of intensity and relationship to vaccination. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Grade 3 irritability/fussiness was defined as crying that could not be comforted/prevented normal activity. Grade 3 loss of appetite was defined as not eating at all. Grade 3 drowsiness was defined as drowsiness that prevented normal activity.Grade 3 fever was defined as axillary temperature above 39.0°C.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: During a 7-day follow-up period (i.e. day of vaccination and six subsequent days) after each vaccination
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 151 | 148
Subjects
  Any Drowsiness | 60 | 56
  Grade 3 Drowsiness | 6 | 3
  Related Drowsiness | 52 | 48
  Any Irritability/fussiness | 76 | 67
  Grade 3 Irritability/fussiness | 13 | 6
  Related Irritability/fussiness | 66 | 60
  Any Loss of appetite | 49 | 46
  Grade 3 Loss of appetite | 5 | 4
  Related Loss of appetite | 46 | 39
  Any Fever | 10 | 10
  Grade 3 Fever | 2 | 3
  Related Fever | 9 | 8

8. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Fever
Description: Any fever was defined as any fever ≥38.0 degrees Celsius (°C) irrespective of intensity and relationship to vaccination. Related was defined as symptoms assessed by the investigator to have a causal relationship to vaccination. Grade 3 fever was defined as fever ≥39.0 °C.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: During a 4-day follow-up period (i.e. day of vaccination and 3 subsequent days) after each vaccination
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 151 | 148
Subjects
  Any Fever | 7 | 8
  Grade 3 Fever | 0 | 1
  Related Fever | 7 | 7

9. Secondary Outcome: Duration of Solicited Local and General Symptoms
Description: Duration was defined as number of days with any grade of local and general symptoms.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: During a 7-day follow-up period (i.e. day of vaccination and six subsequent days) after each vaccination
Population: as for outcome 6
Measure: Median (Full Range); unit: Days
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 64 | 62
Days
  Pain [Dose 1; N=43,44] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 7.0]
  Pain [Dose 2; N=21,11] | 1.0 [1.0 to 5.0] | 1.0 [1.0 to 2.0]
  Redness [Dose 1; N=2,0] | 1.5 [1.0 to 2.0] | 0.0 [0.0 to 0.0]
  Redness [Dose 2; N=0,0] | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event
  Swelling [Dose 1; N=0,1] | NA [NA to NA] — No participants with event | 1.0 [1.0 to 1.0]
  Swelling [Dose 2; N=0,0] | NA [NA to NA] — No participants with event | NA [NA to NA] — No participants with event
  Fever [Dose 1; N=7,8] | 1.0 [1.0 to 6.0] | 1.0 [1.0 to 5.0]
  Fever [Dose 2; N=3,4] | 2.0 [2.0 to 3.0] | 1.5 [1.0 to 3.0]
  Drowsiness [Dose 1; N=56;48] | 1.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Drowsiness [Dose 2; N=22,20] | 2.0 [1.0 to 6.0] | 1.0 [1.0 to 7.0]
  Irritability/fussiness [Dose 1; N=64,62] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 6.0]
  Irritability/fussiness [Dose 2; N=34,27] | 1.0 [1.0 to 6.0] | 2.0 [1.0 to 7.0]
  Loss of appetite [Dose 1; N=41,40] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]
  Loss of appetite [Dose 2; N=17,13] | 2.0 [1.0 to 7.0] | 2.0 [1.0 to 7.0]

10. Secondary Outcome: Number of Subjects Reporting Any Medically Attended Adverse Events (MAEs)
Description: MAEs were defined as adverse events with medically-attended visits that were not routine visits for physical examination or vaccination, such as visits for hospitalization, an emergency room visit, or an otherwise unscheduled visit to or from medical personnel (medical doctor) for any reason. Any was defined as any occurrence of MAE(s). Related was defined as a MAE assessed by the investigator to be causally related to the study vaccination.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: During the entire study period (Day 0 to Day 180)
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 158 | 156
Subjects
  Any MAE(s) | 77 | 89
  Related MAE(s) | 2 | 4

11. Secondary Outcome: Number of Subjects Reporting Any Potential Immune-Mediated Diseases (pIMDs)
Description: pIMDs were defined as a subset of adverse events that included both clearly autoimmune diseases and also other inflammatory and/or neurologic disorders which might or might not have an autoimmune aetiology. Any pIMD was defined as at least one pIMD experienced by the study subject. Related pIMD was defined as a pIMD assessed by the investigator to be causally related to the study vaccination.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: During the entire study period (Day 0 to Day 180)
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 158 | 156
Subjects
  Any pIMD(s) | 0 | 0
  Related pIMD(s) | 0 | 0

12. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Unsolicited Adverse Events (AEs).
Description: An unsolicited AE was defined as an untoward medical occurrence in a patient or clinical investigation subject, temporally associated with use of a medicinal product, whether or not considered related to the medicinal product and reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms. Any was defined as occurrence of any unsolicited symptom regardless of intensity grade or relation to vaccination. Grade 3 was an event that prevented normal activities and related was defined as an unsolicited AE assessed by the investigator to be causally related to the study vaccination
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010
Time Frame: During a 28-day follow-up period (i.e. day of vaccination and 27 subsequent days) after each vaccination
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 158 | 156
Subjects
  Any Unsolicited AEs | 77 | 75
  Grade 3 Unsolicited AEs | 12 | 12
  Related Unsolicited AEs | 11 | 7

13. Secondary Outcome: Number of Subjects Reporting Any and Related Serious Adverse Events (SAEs)
Description: A serious adverse event was defined as any untoward medical occurrence that: resulted in death, was life threatening, required hospitalization or prolongation of hospitalization, resulted in disability/incapacity or was a congenital anomaly/birth defect in the offspring of a study subject. Any was defined as occurrence of any symptom regardless of intensity grade or relation to vaccination and related was an event assessed by the investigator as causally related to the study vaccination.
  Vaccine primed subjects are subjects who had received a total of 2 or more doses of seasonal influenza vaccine since 01 July 2010.
  Vaccine unprimed subjects are subjects who had never received any seasonal influenza vaccine or had received only one dose of seasonal influenza vaccine since 01 July 2010.
Time Frame: During the entire study period (Day 0 - Day 180)
Population: as for outcome 6
Measure: Number; unit: Subjects
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Number analyzed (Participants) | 158 | 156
Subjects
  Any SAEs | 5 | 4
  Related SAEs | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious Adverse Events: From Day 0 to Day 180; Solicited local and general symptoms: During the 7-day (Days 0-6) post-vaccination period; Unsolicited adverse events: During the 28-day (Days 0-27) post-vaccination period.
Description: For the systematically assessed other (non-serious) adverse events, the number of participants at risk included those from Total Vaccinated Cohort who had the symptom sheet completed.
Arm/Group | FluLaval Quadrivalent Group | Fluzone Group
Serious Adverse Events (participants affected / at risk) | 5/158 | 4/156
Other Adverse Events (participants affected / at risk) | 115/158 | 103/156
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | FluLaval Quadrivalent Group (N=158) | Fluzone Group (N=156)
Respiratory syncytial virus infection (Infections and infestations) | 2 | 0
Abscess neck (Infections and infestations) | 0 | 1
Convulsion (Nervous system disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 1
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | FluLaval Quadrivalent Group (N=158) | Fluzone Group (N=156)
Pain (General disorders) | 48/151 | 48/148
Drowsiness (General disorders) | 60/151 | 56/148
Irritability/fussiness (General disorders) | 76/151 | 67/148
Loss of appetite (General disorders) | 49/151 | 46/148
Fever (General disorders) | 10/151 | 10/148 — Assessed during the 7-day (Days 0-6) post-vaccination period
Fever (General disorders) | 7/151 | 8/148 — Assessed duringthe 4-day (Days 0-3) post-vaccination period
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 13
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 13 | 12
Otitis media (Infections and infestations) | 11 | 12
Upper respiratory tract infection (Infections and infestations) | 11 | 11
Nasopharyngitis (Infections and infestations) | 8 | 9
Vomiting (Gastrointestinal disorders) | 9 | 7
Diarrhoea (Gastrointestinal disorders) | 15 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.